CLINICAL TRIAL: NCT06832137
Title: The Efficacy and Safety of CMTS4520 for Chronic Constipation in Adults： A Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: CMTS4520 for Chronic Constipation in Adults
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT-2024CMTS4520-001
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-02

CONDITIONS: Constipation
Keywords: CMTS4520; constipation; randomized controlled trial; dietary fiber; probiotics
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): The patient will receive CMTS4520 (dietary fiber probiotics) capsules daily for 14 days.
  Interventions: Other: CMTS4520 (dietary fiber probiotics)
- Control (Placebo Comparator): The patient will receive placebo of equal capsules daily for 14 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: CMTS4520 (dietary fiber probiotics) — CMTS4520 is a synbiotic formulation containing a standardized ratio of plant-derived prebiotics and clinically validated probiotic strains. Participants will receive 2 weeks of CMTS4520 daily for chronic constipation.
  Arms: Treatment
Other: Placebo — Capsules with matching volume and consistent appearance to CMTS4520.
  Arms: Control

SUMMARY:
This is a randomized controlled trial to explore the efficacy and safety of CMTS4520 (Dietary Fiber Probiotics) for patients with chronic constipation.

DETAILED DESCRIPTION:
At least 100 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. They will be randomly assigned to the CMTS4520 group (dietary fiber probiotics capsules) and the control group (placebo). Data of demographic characteristics, intestinal symptoms, medicine treatment usage and clinical outcomes will be collected. After treatment, they will enter the follow-up period for efficacy and safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

-

Meet all of the following inclusion criteria :

1. Voluntary sign informed consent, age 18-70 years old (including the threshold), male and female.
2. For subjects diagnosed with chronic constipation, the duration of the disease is at least 6 months, and meet the following criteria:

   1. Frequency of spontaneous defecation <3 times/week (spontaneous defecation refers to spontaneous defecation without the aid of remedial purgatives or manual assistance).
   2. Dry and hard stool: More than a quarter of the stool is type 1 or 2 on the Bristol Fecal Trait Scale.
3. The subject or his/her legal representative has given informed consent, is fully aware of the purpose of the study, is able to communicate well with the investigator, and is able to understand and comply with the requirements of the study.

Exclusion Criteria:

-

All exclusion criteria below are not met:

1. Participants with outlet obstruction constipation, such as rectal mucosal prolapse.
2. Participants with a history of intestinal resection.
3. Participants with intestinal stenosis caused by organic lesions of the digestive tract (e.g., tumor, inflammation, anal fissures, Crohn's disease, ulcerative colitis, radiation enteritis, intestinal adhesions, intestinal tuberculosis) as confirmed by colonoscopy within the past 24 months.
4. Participants with constipation secondary to systemic diseases affecting the digestive tract, including:

   1. Neurological diseases (e.g., Parkinson's disease, spinal cord injury, multiple sclerosis).
   2. Muscle diseases (e.g., amyloidosis, dermatomyositis).
   3. Psychiatric disorders or severe mood disorders (e.g., A Hospital Anxiety and Depression Scale score ≥15).
   4. Opioid-induced constipation.
   5. Poorly controlled metabolic diseases (e.g., thyroid dysfunction) or metabolic diseases with gastrointestinal complications (e.g., gastrointestinal autonomic dysfunction, diabetic gastroparesis).
5. Have a history of major surgery or severe trauma within 3 months and have not fully recovered.
6. Participants with any of the following cardiac abnormalities:

   1. New York Heart Association (NYHA) Class III or higher heart failure.
   2. Myocardial infarction or unstable angina within the past 6 months.
   3. Prolonged QTc interval on electrocardiogram (≥450ms for males, ≥470ms for females).
   4. Atrial arrhythmias that cannot be stably controlled by drugs and ventricular arrhythmias requiring pharmacological control (including grade 2 or higher atrioventricular block).
7. Participants with poor lung function, as assessed by the investigator, that may impact study treatment, such as acute chronic obstructive pulmonary disease(COPD) or those requring long-term oral, intravenous corticosteroids (excluding inhalant/spray formulations).
8. Uncontrolled immune diseases requring long-term systemic corticosteroid use (excluding topical use).
9. Participants with reproductive system disorders that may cause abdominal pain (e.g., ovarian cysts, endometriosis, primary dysmenorrhea).
10. Participants with significant laboratory abnormalities that, in the investigator's judgment, may affect safety or study completion, including:

    1. Hemoglobin <100g/L.
    2. Serum creatinine ≥1.5 times the upper limit of normal (ULN).
    3. Abnormal liver function (AST>1.5×ULN, ALT>1.5×ULN or total bilirubin >1.5×ULN).
    4. Clinically significant abnormalitieshe in routine stool tests or fecal occult blood indicating gastrointestinal lesions.
11. Participants with active hepatitis (requiring or undergoing long-term treatment), HIV, or active tuberculosis.
12. Participants with a history of drug or alcohol abuse (defined as consuming more than 14 standard drinks peer week: 1 standard drink= 360mL of beer, 45mL of 40% spirits, or 150mL of wine) or substance abuse.
13. Participants with known allergies or intolerances to the investigational drug, similar drugs or excipients.
14. Participants who have used anti-infective drugs (antibiotics, antifungals, antivirals) within 14 days prior to enrollment or require anti-infective treatment at the time of enrollment evaluation.
15. Participants who have used drugs or foods that regulate intestinal microbiota (e.g., bifidobacterium, probiotics, prebiotics, fermented milk, yogurt) within 2 weeks prior to screening or during the study.
16. Participants who have undergone hydrotherapy for bowel cleansing within one month prior to treatment.
17. Women who are pregnant, breastfeeding, or unwilling to use effective contraception for 3 months after the last dose of the study drug.
18. Participants who have participated in drug intervention clinical trials within 1 month prior to enrollment.
19. Any other condition that, in the investigator's judgment, makes the participant unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
The clinical response rate after treatment | One-week post-CMTS4520 administration，Two-week post-CMTS4520 administration，Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  A clinical response was defined as a patient achieving complete spontaneous bowel movement (CSBM) at least 50% of the time after receiving CMTS4520. CSBM was defined as the number of spontaneous defecation with complete exhaust feeling without taking remedial purgative or manual assistance.

SECONDARY OUTCOMES:
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | Two-week post-CMTS4520 adminiatration, Four-week post-CMTS4520 administration，Eight-week post-CMTS4520 administration
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).
The weekly usage rate of assisted defecation drugs. | One-week post-CMTS4520 administraion，Two-week post-CMTS4520 administraion, Four-week post-CMTS4520 administraion，Eight-week post-CMTS4520 administraion
  Percentage of days per week after CMTS4520 that assisted defecation drugs were used, which was compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases,The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lembo AJ, Kurtz CB, Macdougall JE, Lavins BJ, Currie MG, Fitch DA, Jeglinski BI, Johnston JM. Efficacy of linaclotide for patients with chronic constipation. Gastroenterology. 2010 Mar;138(3):886-95.e1. doi: 10.1053/j.gastro.2009.12.050. Epub 2010 Jan 4. PMID 20045700
- [Background] Schoenfeld P, Lacy BE, Chey WD, Lembo AJ, Kurtz CB, Reasner DS, Bochenek W, Tripp K, Currie MG, Fox SM, Blakesley RE, O'Dea CR, Omniewski ND, Hall ML. Low-Dose Linaclotide (72 mug) for Chronic Idiopathic Constipation: A 12-Week, Randomized, Double-Blind, Placebo-Controlled Trial. Am J Gastroenterol. 2018 Jan;113(1):105-114. doi: 10.1038/ajg.2017.230. Epub 2017 Aug 22. PMID 29091082
- [Background] Khalif IL, Quigley EM, Konovitch EA, Maximova ID. Alterations in the colonic flora and intestinal permeability and evidence of immune activation in chronic constipation. Dig Liver Dis. 2005 Nov;37(11):838-49. doi: 10.1016/j.dld.2005.06.008. Epub 2005 Oct 5. PMID 16169298
- [Background] Korolkiewicz PK. Commentary on: "Does caffeine enhance bowel recovery after elective colorectal resection? A prospective double-blinded randomized clinical trial" Tech Coloproctol. 2021 Apr 26. doi: 10.1007/s10151-021-02450-7. Tech Coloproctol. 2021 Sep;25(9):1095-1096. doi: 10.1007/s10151-021-02489-6. Epub 2021 Jun 25. No abstract available. PMID 34170420
- [Background] Waitzberg DL, Logullo LC, Bittencourt AF, Torrinhas RS, Shiroma GM, Paulino NP, Teixeira-da-Silva ML. Effect of synbiotic in constipated adult women - a randomized, double-blind, placebo-controlled study of clinical response. Clin Nutr. 2013 Feb;32(1):27-33. doi: 10.1016/j.clnu.2012.08.010. Epub 2012 Aug 23. PMID 22959620
- [Background] Fosch SE, Ficoseco CA, Marchesi A, Cocucci S, Nader-Macias MEF, Perazzi BE. Contraception: Influence on Vaginal Microbiota and Identification of Vaginal Lactobacilli Using MALDI-TOF MS and 16S rDNA Sequencing. Open Microbiol J. 2018 Jun 29;12:218-229. doi: 10.2174/1874285801812010218. eCollection 2018. PMID 30069261
- [Background] Vazquez Roque M, Bouras EP. Epidemiology and management of chronic constipation in elderly patients. Clin Interv Aging. 2015 Jun 2;10:919-30. doi: 10.2147/CIA.S54304. eCollection 2015. PMID 26082622
- [Background] Gallegos-Orozco JF, Foxx-Orenstein AE, Sterler SM, Stoa JM. Chronic constipation in the elderly. Am J Gastroenterol. 2012 Jan;107(1):18-25; quiz 26. doi: 10.1038/ajg.2011.349. Epub 2011 Oct 11. PMID 21989145
- [Background] Fleming V, Wade WE. A review of laxative therapies for treatment of chronic constipation in older adults. Am J Geriatr Pharmacother. 2010 Dec;8(6):514-50. doi: 10.1016/S1543-5946(10)80003-0. PMID 21356503
- [Background] Zhao YF, Ma XQ, Wang R, Yan XY, Li ZS, Zou DW, He J. Epidemiology of functional constipation and comparison with constipation-predominant irritable bowel syndrome: the Systematic Investigation of Gastrointestinal Diseases in China (SILC). Aliment Pharmacol Ther. 2011 Oct;34(8):1020-9. doi: 10.1111/j.1365-2036.2011.04809.x. Epub 2011 Aug 17. PMID 21848795
- [Background] Chu H, Zhong L, Li H, Zhang X, Zhang J, Hou X. Epidemiology characteristics of constipation for general population, pediatric population, and elderly population in china. Gastroenterol Res Pract. 2014;2014:532734. doi: 10.1155/2014/532734. Epub 2014 Oct 16. PMID 25386187
- [Background] Long Y, Huang Z, Deng Y, Chu H, Zheng X, Yang J, Zhu Y, Fried M, Fox M, Dai N. Prevalence and risk factors for functional bowel disorders in South China: a population based study using the Rome III criteria. Neurogastroenterol Motil. 2017 Jan;29(1). doi: 10.1111/nmo.12897. Epub 2016 Jul 14. PMID 27412422
- [Background] Pare P, Ferrazzi S, Thompson WG, Irvine EJ, Rance L. An epidemiological survey of constipation in canada: definitions, rates, demographics, and predictors of health care seeking. Am J Gastroenterol. 2001 Nov;96(11):3130-7. doi: 10.1111/j.1572-0241.2001.05259.x. PMID 11721760